CLINICAL TRIAL: NCT06866158
Title: Single-arm Open-label Clinical Trial: Autologous Dendritic Cells and Lymphocytes in Type 2 Diabetes Mellitus With Albuminuria
Brief Title: Autologous Dendritic Cell as Adjunct Therapy for Diabetic Kidney Disease
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PT. JES Kasih Nusantara Sejahterah (Industry)
Collaborators: Rumah Sakit Pusat Angkatan Darat Gatot Soebroto (Other); Universitas Prima Indonesia (Unknown); Universitas Pertahanan Indonesia (Unknown)
Responsible Party: Principal Investigator, dr. Jonny, Sp.PD-KGH, M.Kes, M.M, DCN, Principal Investigator, Rumah Sakit Pusat Angkatan Darat Gatot Soebroto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-DKD-P01-ID
Record Dates: First submitted 2025-02-22; First posted 2025-03-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Kidney Disease (DKD)
Keywords: Dendritic Cell; Immunotherapy; Diabetic Kidney Disease; Cellular Therapy; Autologous
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Intervention Model Description: All subjects that fulfilled the enrollment criteria were given a single dose of autologous DC therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous DCL (Experimental)
  Interventions: Biological: Dendritic cell immunotherapy

INTERVENTIONS:
Biological: Dendritic cell immunotherapy — DCL (Dendritic Cells+Lymphocytes) previously matured with S-Protein of SARS-CoV-2. The number of cells given depends on individual yields.
  Other Names: Immunotherapy Nusantara

SUMMARY:
The goal of this single-arm, open-label clinical trial is to evaluate the effects of subcutaneous autologous dendritic cell (DC) and lymphocyte administration on albuminuria and endothelial dysfunction in Type 2 Diabetes Mellitus (T2DM) patients with Diabetic Kidney Disease (DKD). The main questions it aims to answer are:

* Does autologous DC immunotherapy reduce urine albumin-creatinine ratio (UACR) in DKD patients?
* What are the underlying mechanisms (modulation of inflammation, endothelial dysfunction, angiogenesis, fibrosis, and structural changes) through which DC immunotherapy reduces UACR in DKD patients?

Participants will:

* Undergo collection of autologous dendritic cells, which will be matured ex vivo using SARS-CoV-2 S protein.
* Receive a single subcutaneous injection consisting of matured dendritic cells and lymphocyte reinfusion.
* Have UACR measured at baseline and at weeks 1, 2, 3, and 4 post-immunotherapy.
* Undergo assessments of other laboratory parameters and kidney imaging (ultrasonography and/or magnetic resonance imaging) at baseline and week 4 post-treatment.
* What is the effect of autologous DC immunotherapy on knee OA, assessed by radiographic changes (x-ray) and patient-reported outcomes (WOMAC score)?

Additionally, a subgroup of subjects who had neuropathy as comorbidity will be assessed using Electromyography (EMG) and the Toronto Clinical Neuropathy Scale (TCNS). These assessments aimed to determine the impact of the intervention on peripheral nerve function, clinical neuropathy symptoms over the study period. Another subgroup of subjects who had knee osteoarthritis will be assessed their knee x-ray and Western Ontario and McMaster Universities osteoarthritis index (WOMAC) score. These assessments aimed to determine the impact of the intervention on knee anatomic structure, function, and pain.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over 18 years old
2. Understands and agrees to comply with study procedures by providing written informed consent.
3. In the investigator's judgment, the subject is able and willing to comply with study procedures.
4. In the investigator's judgment, the subject is in generally good physical and mental health. This includes the following factors:

   * Age > 65 years
   * Mild to moderate obesity (BMI 30 to 40)
   * Controlled hypertension with medication
   * Controlled hyperlipidemia with medication
   * Mild chronic lung disease
   * Previously diagnosed with cancer and in remission for at least 1 year
5. Meets the diagnostic criteria for Type 2 Diabetes Mellitus (DM) according to Indonesia's Endocrinology Society (PERKENI) 2021.
6. eGFR ≥ 30 mL/min/1.73 m².
7. Urinary albumin-creatinine ratio (UACR) ≥ 30 mg/g.

Exclusion Criteria:

1. Receiving immunosuppressive treatments such as corticosteroids, hydroxychloroquine, methotrexate, cyclophosphamide, and others within the last 4 weeks.
2. Known to have other kidney diseases (e.g., polycystic kidney disease, lupus nephritis, ANCA-associated vasculitis, etc.).
3. Known to have other conditions that can cause albuminuria (e.g., myeloma, rhabdomyolysis, paroxysmal nocturnal hemoglobinuria, orthostatic albuminuria, etc.).
4. Diagnosed with other types of diabetes (Type 1 DM, gestational DM, or other forms of DM).
5. Positive pregnancy test.
6. Known to have immunodeficiency diseases such as human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV); no blood testing required.
7. Requires oxygen supplementation.
8. Diagnosed with invasive cancer and currently receiving anti-cancer therapy, except for hormonal therapy for breast or prostate cancer.
9. History of thromboembolism or a genetic predisposition to thromboembolism, or currently on anti-thromboembolic therapy other than low-dose aspirin.
10. Physical or mental disabilities preventing normal daily activities.
11. In the investigator's judgment, any illness or medical condition that may hinder the subject's participation, including acute, subacute, intermittent, or chronic diseases that could place the subject at risk of injury, prevent compliance with the study protocol, or interfere with study assessments.
12. Measurable parameters include:

    * Severe obesity: BMI > 40
    * Uncontrolled hypertension: systolic >180 mmHg, diastolic >100 mmHg
13. Unwilling to sign the written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2026-08-05 (Estimated)

PRIMARY OUTCOMES:
Change in Urine Albumin-Creatinine Ratio (UACR) from Baseline | From baseline to 4 weeks after treament
  UACR were evaluated at a total 5 time points: baseline, week 1, 2, 3, and 4.

SECONDARY OUTCOMES:
Change in Estimated Glomerular Filtration Rate | From baseline to 4 weeks after treament
  Estimated glomerular filtration rate (eGFR) calculated from serum creatinine using the CKD-EPI equation.
Change in Angiogenesis Biomarker | From baseline to 4 weeks after treament
  An angiogenesis biomarker, vascular endothelial growth factor (VEGF) were evaluated at baseline and 4 weeks post-treatment. With measurements expressed in pg/mL.
Change in Interleukin-6 | From baseline to 4 weeks after treament
  Interleukin-6 (IL-6), an inflammatory biomarker, was evaluated at both baseline and 4 weeks post-treatment. With measurements expressed in pg/mL.
Change in tumor necrosis factor-α | From baseline to 4 weeks after treament
  Tumor necrosis factor-α (TNF-α), an inflammatory biomarker, was evaluated at both baseline and 4 weeks post-treatment. With measurements expressed in pg/mL.
Change in interleukin-10 | From baseline to 4 weeks after treament
  Interleukin-10 (IL-10), an inflammatory biomarker, was evaluated at both baseline and 4 weeks post-treatment. With measurements expressed in pg/mL.
Change in transforming growth factor-β | From baseline to 4 weeks after treament
  Transforming growth factor-β (TGF-β), an endothelial biomarkers, were evaluated at baseline and 4 weeks post-treatment. With measurements expressed in pg/mL.
Change in matrix metalloproteinase-9 | From baseline to 4 weeks after treament
  Change in matrix metalloproteinase-9 (MMP-9), an endothelial biomarkers, were evaluated at baseline and 4 weeks post-treatment. With measurements expressed in ng/mL.
Change in endhotelin | From baseline to 4 weeks after treament
  Endhotelin, an endothelial biomarkers, were evaluated at baseline and 4 weeks post-treatment. With measurements expressed in pg/mL.
Change in intercellular adhesion molecule | From baseline to 4 weeks after treament
  Change in intercellular adhesion molecule (ICAM), an endothelial biomarkers, were evaluated at baseline and 4 weeks post-treatment. With measurements expressed in ng/mL.
Change in vascular cell adhesion protein | From baseline to 4 weeks after treament
  Change in vascular cell adhesion protein (VCAM), an endothelial biomarkers, were evaluated at baseline and 4 weeks post-treatment. With measurements expressed in ng/mL.
Change in kidney perfusion | From baseline to 4 weeks after treament
  Doppler Ultrasonography (Doppler USG) of the kidneys were performed at baseline and 4 weeks post-treatment.
Change in kidney tissue and function | From baseline to 4 weeks after treament
  Magnetic Resonance Imaging Diffusion Weighted Imaging (MRI DWI) of the kidneys were performed at baseline and 4 weeks post-treatment.
Change in kidney tissue and function | From baseline to 4 weeks after treament
  Magnetic Resonance Imaging Diffusion Tensor Imaging (MRI DTI) of the kidneys were performed at baseline and 4 weeks post-treatment.

OTHER OUTCOMES:
Change in Nerve Conduction Velocity | From baseline to 4 weeks after treament
  Changes in Nerve Conduction Velocity (m/s) as measured by Electromyography were conducted only on a subgroup of patients who had Neuropathy as a comorbidity and were assessed at two time points: baseline and 4 weeks post-treatment.
Change in Toronto Clinical Neuropathy Score | From baseline to 4 weeks after treament
  Changes in Toronto Clinical Neuropathy Score (TCNS) were conducted only on a subgroup of patients who had Neuropathy as a comorbidity and were assessed at two time points: baseline and 4 weeks post-treatment.This scale is used to assess the severity of diabetic peripheral neuropathy. The score ranges from 0 to 15, with higher scores indicating worse neuropathy. It evaluates various clinical signs, such as the presence of symptoms like pain, numbness, and weakness, along with physical examination findings like ankle reflexes and vibration sensation. A higher score suggests more severe neuropathy and a worse outcome for the patient.
Knee X-ray | Baseline and 4 weeks after intervention
  Knee X-ray done on both knee and graded using Kellgren-Lawrence grading system
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Baseline to 4 weeks after intervention
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a self-administered questionnaire for assessing pain, stiffness, and physical function in individuals with osteoarthritis of the hip or knee. The WOMAC is a 24-item tool that includes 5 questions on pain, 2 on stiffness, and 17 on physical function, with higher scores indicating worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: dr Jonny, Sp.PD-KGH, M.Kes, M.M, DCN, Principal Investigator — Gatot Soebroto Central Army Hospital
Locations (1):
- Gatot Soebroto Central Army Hospital, Jakarta Pusat, DKI Jakarta - Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Only individual participant data (IPD) underlying the results presented in the publication will be shared.

REFERENCES:
- [Background] Jonny J, Sitepu EC, Lister INE, Chiuman L, Putranto TA. The Potential of Anti-Inflammatory DC Immunotherapy in Improving Proteinuria in Type 2 Diabetes Mellitus. Vaccines (Basel). 2024 Aug 27;12(9):972. doi: 10.3390/vaccines12090972. PMID 39340004
- [Result] Setiawan E, Ginting CN, Jonny J, Hernowo BA, Putranto TA. Clinical Trial: Effect of Autologous Dendritic Cell Administration on Improving Neuropathy Symptoms and Inflammatory Biomarkers in Diabetic Neuropathy. Curr Issues Mol Biol. 2024 Dec 20;46(12):14366-14380. doi: 10.3390/cimb46120861. PMID 39727989
- [Result] Dimu PS, Icksan AG, Farhat, Jonny, Hernowo BA, Putranto TA. Clinical Trial of Autologous Dendritic Cell Administration Effect on Water Molecule Diffusion and Anti-Inflammatory Biomarkers in Diabetic Kidney Disease. Curr Issues Mol Biol. 2024 Dec 4;46(12):13767-13779. doi: 10.3390/cimb46120822. PMID 39727950
- [Result] Jonny, Sitepu EC, Hernowo BA, Chiuman L, Lister INE, Putranto TA. Open-Label Clinical Trial on the Impact of Autologous Dendritic Cell Therapy on Albuminuria and Inflammatory Biomarkers (Interleukin-6, Interleukin-10, Tumor Necrosis Factor alpha) in Diabetic Kidney Disease (DKD). Curr Issues Mol Biol. 2024 Dec 2;46(12):13662-13674. doi: 10.3390/cimb46120816. PMID 39727944
- [Result] Yana ML, Sitepu EC, Jonny, Chiuman L, Lister INE, Putranto TA. The Effect of Autologous Dendritic Cell Immunotherapy on Kidney Function and Endothelial Dysfunction of Patients with Diabetic Kidney Disease (DKD): An Open Label Clinical Trial. Curr Issues Mol Biol. 2025 Jan 6;47(1):31. doi: 10.3390/cimb47010031. PMID 39852146